CLINICAL TRIAL: NCT06125977
Title: The Impact of Non-Exudative Type 1 Macular Neovascularization (MNV) on Age-related Macular Degeneration (AMD) Progression
Brief Title: Impact of Non-Exudative Type 1 MNV on AMD Progression
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Monika Fleckenstein, Professor, University of Utah
Other Study IDs: IRB_00151913; 1R01EY033365-01A1 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-11-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Age-Related Macular Degeneration; Neovascularization, Choroidal
Keywords: Non-exudative type 1 macular neovascularization (MNV)
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Intermediate AMD group, Original Cohort
- Cohort 2: Atrophic AMD and/or previous treatment group, Extended Cohort

SUMMARY:
The overall goal of the proposed research project is to provide evidence that a specific subtype of neovascularization that may develop in eyes with age-related macular degeneration (AMD) prevents vision loss.

This concept challenges the current view that the development of neovascularizations in AMD represents a harmful event in general. Notably, before the era of anti-vascular endothelial growths factor (VEGF) therapy, destruction and surgical removal of neovascular membranes have been tested as treatment options for neovascular AMD.

This research project aims to substantiate the hypothesis that type 1 macular neovascularization (MNV) is intrinsically protective, in sense of a positive response to the degenerative processes in AMD. This concept has actually been proposed by pathologists decades ago but has not been systematically investigated in vivo.

With the immense advances in retinal imaging, 'sub-clinical', non-exudative type 1 MNVs that are located beneath the retinal pigment epithelium (RPE) can now be detected non-invasively and characterized in vivo. There is currently a growing body of evidence that photoreceptor and RPE degeneration is indeed slowed down in eyes exhibiting type 1 MNV. However, the proof of a direct protective effect of non-exudative type 1 MNV on visual function in AMD is lacking.

Here, the aim is to demonstrate relative preservation of function along with preserved structure in the immediate vicinity of type 1 MNV, while there is progressive loss of sensitivity and degeneration in the surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 50 years and older of all ethnicities.
2. AMD in at least one eye (study eye).
3. Type 1 macular neovascularization (MNV) in the study eye (to be confirmed by UREAD Reading Center at the Screening and Baseline Visit):

   1. Localized presence of a dense vascular network between Bruch's membrane and retinal pigment epithelium (RPE) on optical coherence tomography angiography (OCT-A) and a double-layer / shallow irregular RPE elevation (SIRE) sign on structural OCT.
   2. MNV lesion does not exceed the image frame of the 9x9 OCT-A scan.
4. Sufficiently clear ocular media, adequate pupillary dilation, and adequate fixation to permit quality fundus imaging and fundus-controlled perimetry (FCP) testing.
5. Ability to comply with study protocol timelines.

Exclusion Criteria:

Intermediate AMD group (original cohort): Exclusion criteria 1. - 11. apply. Atrophic AMD and/or previous treatment group (extended cohort): Exclusion criteria 4. - 11. apply.

1. Atrophy in the study eye defined as:

   * Complete RPE and outer retinal atrophy (cRORA) on OCT with homogeneous choroidal hypertransmission
   * Absence of the RPE band measuring > 250 microns
   * Evidence of overlying photoreceptor degeneration whose features include outer nuclear layer thinning, external limiting membrane loss, and ellipsoid zone or interdigitation zone loss
2. Signs of exudation in the study eye requiring therapeutic intervention at the discretion of the investigator; NOTE: minimally exudative lesions in the study eye that do not require therapeutic interventions are no exclusion criterion.
3. Any history of treatment of exudative MNV in the study eye (e.g. type 1, type 2, mixed, polypoidal choroidal vasculopathy, and retinal angiomatous proliferation); NOTE: Non-exudative or minimally exudative type 1 MNV in the study eye, that does not require therapeutic intervention at the discretion of the investigator, is NOT and exclusion criterion; non-exudative or exudative MNV in the fellow eye is not an exclusion criterion. Fellow-eyes may receive treatment of exudative MNV as part of clinical care.
4. Any disease/disorder other than AMD in the study eye at the time of inclusion (e.g. monogenic retinal diseases, diabetic retinopathy, retinal detachment, previous retinal surgeries, myopic degeneration), uncontrolled glaucoma with IP of higher than 30 mmHg (despite current pharmacological or non-pharmacological treatment) and uveitis.
5. History of central retinal laser treatment, including photodynamic therapy (PDT) and subthreshold laser treatment for AMD in the study eye.
6. Cataract surgery in the study eye within the last three months prior to enrollment. YAG capsulotomy in the study eye within the last 2 weeks prior to enrollment.
7. Current or previous participation in clinical trials investigating drugs or supplements in AMD (except vitamins and minerals), if, in the opinion of the investigator, this affects the outcome of the study.
8. Current or previous participation (less than 3 months from termination of participation) in clinical trials investigating drugs or supplements in diseases other than AMD, if, in the opinion of the investigator, this affects the outcome of the study.
9. Any concurrent ocular condition in the study eye (e.g. cataracts) that, in the opinion of the investigator, requires medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition or, if allow to progress untreated, could likely contribute to loss of at least two Snellen equivalent lines of best-corrected visual acuity during the study period.
10. Concomitant diseases that in the opinion of the investigator would make adherence to the examination schedule difficult of unlikely (e.g. personality disorder, chronic alcoholism, Alzheimer's Disease, drug abuse).
11. Evidence of significantly uncontrolled concomitant diseases at the discretion of the investigator (e.g. cardiovascular, neurological, pulmonary, renal, hepatic, endocrine gastrointestinal disorder).

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with AMD.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Mean change in mesopic retinal sensitivity assessed by Fundus-controlled Perimetry (FCP). | At months 36 from baseline.
  This sensitivity change will be compared between (I) retinal areas colocalizing with non-exudative type 1 MNV (test-point group I) and (II) retinal areas without evidence of MNV (testpoint group II).

SECONDARY OUTCOMES:
Changes over time of qualitative and quantitative structural biomarkers for disease progression. | At months 36 from baseline.
  These changes will be compared between (I) retinal areas co-localizing with non-exudative type 1 MNV and (II) retinal areas without evidence of MNV.
Mean change over time in dark-adapted retinal sensitivity assessed by Fundus-controlled Perimetry (FCP). | At months 36 from baseline.
  This sensitivity change will be compared between (I) retinal areas colocalizing with non-exudative type 1 MNV (test-point group I) and (II) retinal areas without evidence of MNV (testpoint group II).

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fleckenstein, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States